CLINICAL TRIAL: NCT03493048
Title: Cetuximab Plus FOLFOXIRI vs Cetuximab Plus FOLFOX in Patients With Initially Unresectable Colorectal Liver Metastasis
Brief Title: Cetuximab Plus FOLFOXIRI vs Cetuximab Plus FOLFOX For CRCLM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERBIRINOX-CRCLM
Record Dates: First submitted 2018-03-27; First posted 2018-04-10 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Liver Metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Cetuximab; Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cetuximab Plus FOLFOXIRI (Experimental): Cetuximab Plus FOLFOXIRI Patients will receive Cetuximab Plus FOLFOXIRI every 14 days: Cetuximab 500mg/m2 ivd over 90 minutes on Day 1; Oxaliplatin 85 mg/m2 ivd over 3 hours on Day 1; Irinotecan 130 mg/m2 ivd over 90 minutes on Day 1; Leucovorin (l-LV) 200mg/m2 ivd over 2 hours on Day 1; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion on Day 1.
  Interventions: Drug: Irinotecan; Drug: Cetuximab; Drug: 5-fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin
- Cetuximab Plus FOLFOX (Active Comparator): Patients will receive Cetuximab Plus FOLFOX every 14 days: Cetuximab 500mg/m2 ivd over 90 minutes on Day 1; Oxaliplatin 85 mg/m2 ivd over 3 hours on Day 1; Leucovorin (l-LV) 200mg/m2 ivd over 2 hours on Day 1; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion on Day 1.
  Interventions: Drug: Cetuximab; Drug: 5-fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 130 mg/m²
  Other Names: CPT-11
  Arms: Cetuximab Plus FOLFOXIRI
Drug: Cetuximab — Cetuximab, iv, 500mg/m2
  Other Names: Erbitux
Drug: 5-fluorouracil — 5-FU 2400 mg/m² cont. inf.
  Other Names: 5-FU
Drug: Oxaliplatin — oxaliplatin 85 mg/m²
  Other Names: L-OHP
Drug: Leucovorin — leucovorin 200 mg/m²
  Other Names: FOLINIC ACID

SUMMARY:
The aim of the trial is to optimize response rates and rates of secondary resections of metastases in patients with initially non-resectable metastatic colorectal cancer Liver Metastasis of RAS wildtype. The patients will be treated in two therapy groups:

Experimental arm A: Chemotherapy with FOLFOXIRI + Cetuximab Standard arm B: Chemotherapy with FOLFOX + Cetuximab

DETAILED DESCRIPTION:
We intend to carry out a randomized controlled clinical study of cetuximab plus FOLFOXIRI regimen versus cetuximab plus FOLFOX regimen in the first-line treatment of patients with initially unresectable CRLM, to answer the question of whether cetuximab plus FOLFOXIRI regimen can improve the overall ORR, surgical resection rate and OS compared with cetuximab plus FOLFOX regimen in patients with previously untreated, initially unresectable CRLM patients.

ELIGIBILITY:
Inclusion criteria

1. Age ≥ 18 years and ≤ 70 years.
2. Histologically confirmed colorectal adenocarcinoma.
3. Liver metastasis confirmed by imaging or pathology.
4. The multidisciplinary team (MDT) determines that the liver metastases are unresectable, which is specifically defined as ① metastatic lesions ≥ 5; ② ineligible for R0 resection; ③ expected insufficient residual liver volume after resection; ④ unable to preserve all three hepatic veins after resection, unable to ensure that the blood flow and bile ducts of the residual liver into and out of the liver could be preserved, and unable to preserve the adjacent two liver segments. Patients who meet any of the above criteria can be determined as having initially unresectable liver metastases.
5. Patients with wild-type RAS.
6. No prior treatment for liver metastases, including chemotherapy, surgery, radiotherapy, transcatheter arterial chemoembolization (TACE), and targeted therapy.
7. Absence of extrahepatic metastasis confirmed by CT, MRI or PET/CT (if necessary) (enrollment can be considered if there is a lung or lymph node lesion less than 10 mm, which is difficult to determine metastases).
8. Normal hematologic function (platelets > 90 × 109/L; leukocytes > 3 × 109/L; neutrophils > 1.5 × 109/L).
9. Serum bilirubin ≤ 1.5 times the upper limit of normal (ULN) and transaminases ≤ 5 times ULN.
10. No ascites, normal coagulation function, albumin ≥ 35 g/L.
11. Liver function: Child-Push score: Class A
12. Serum creatinine < ULN, or calculated creatinine clearance > 50 ml/min (using the Cockcroft-Gault formula).
13. ECOG score 0-1.
14. Life expectancy > 3 months.
15. Sign written informed consent.
16. Willing and able to be followed up until death or end of study or study termination.

Exclusion criteria:

1. Presence of any extrahepatic metastasis and/or primary tumor that cannot be resected with radical surgery.
2. Serious arterial embolism or ascites.
3. Have bleeding tendency or coagulation disorder.
4. Have hypertensive risk or hypertensive encephalopathy.
5. Serious uncontrolled systemic complications such as infection or diabetes.
6. Clinically significant cardiovascular disease such as cerebrovascular accident (within 6 months prior to enrollment), myocardial infarction (within 6 months prior to enrollment), uncontrolled hypertension despite appropriate medical treatment. Unstable angina, congestive heart failure (NYHA class 2-4), cardiac arrhythmia requiring medication.
7. History or physical evidence of central nervous system disease (e.g., primary brain tumor, epilepsy uncontrolled by standard of care, any history of brain metastases or stroke).
8. History of other malignancies (except basal cell carcinoma of the skin and/or carcinoma in situ of the cervix after radical surgery) within the past 5 years.
9. Treatment with any ongoing investigational drug within the last 28 days prior to the study.
10. Any residual toxicity from prior chemotherapy (except alopecia), such as peripheral neuropathy ≥ NCI CTC v4.03 Grade 2, will not be considered for oxaliplatin-containing regimen.
11. Hypersensitivity to any drug in the study.
12. Pregnant and lactating women.
13. Women of childbearing age (< 2 years after menstruation) or men of childbearing potential who are not using or refuse to use effective non-hormonal contraception (intrauterine contraceptive ring, barrier contraceptives combined with spermicidal gel, or surgical sterilization).
14. Unable or unwilling to comply with the study protocol.
15. Patients with any other diseases, dysfunction caused by metastatic lesions, or suspected disease found by physical examination, indicating possible contraindications to the use of the investigational drug or putting the patients at high risk of treatment-related complications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | assessed up to 12 months
  Partial response (PR) plus complete response (CR)): assessed by the investigator using RECIST v1.1 criteria

SECONDARY OUTCOMES:
Depth of Response | Each follow up visit, assessed up to 12 months
  The investigator assesses DpR by measuring the ratio of maximum tumor regression to baseline tumor, and calculates the median value
R0 Resection Rate | Each follow up visit, assessed up to 12 months
  Defined as the proportion of patients who achieve complete resection after treatment with cetuximab plus FOLFOXIRI regimen or cetuximab plus FOLFOX regimen according to the study protocol
Early Tumor Shrinkage | Each follow up visit, assessed up to 12 months
  Target lesion reduction of a least 20% from the nadir following 4 treatment courses assessed using the RECIST version 1.1 criteria
Progression-Free Survival | Each follow up visit, assessed up to 60 months
  Assessed by the investigator using RECIST v1.1, defined as the time from the start of study treatment to disease progression, or relapse after resection of liver metastases, or death due to any cause.
Overall Survival | Each follow up visit, assessed up to 60 months
  Defined as the time from the start of study treatment to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Yuhong Li, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang DS, Ren C, Li SS, Fong WP, Wu XJ, Xiao J, Li BK, Zheng Y, Ding PR, Chen G, Qiu MZ, Wang ZQ, Wang FH, Luo HY, Wang F, Wang XZ, Wang LY, Xie DJ, Chen T, Li LR, Lu ZH, Zhai XH, Liu TS, Yuan Y, Chen JQ, Tan Q, Pan ZZ, Wan DS, Zhang R, Yuan YF, Xu RH, Li YH. Cetuximab plus FOLFOXIRI versus cetuximab plus FOLFOX as conversion regimen in RAS/BRAF wild-type patients with initially unresectable colorectal liver metastases (TRICE trial): A randomized controlled trial. PLoS Med. 2024 May 10;21(5):e1004389. doi: 10.1371/journal.pmed.1004389. eCollection 2024 May. PMID 38728364